CLINICAL TRIAL: NCT05715593
Title: The Effectiveness of a Health Education Intervention to Reduce Anxiety in Quarantined COVID-19 Patients: A Randomized Controlled Trial
Brief Title: The Effectiveness of a Health Education Intervention to Reduce Anxiety in Quarantined COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Imen Zemni, Medical doctor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMONASTIR1
Record Dates: First submitted 2023-02-03; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Health Education, COVID-19, Quarantine, Anxiety, Pandemic
MeSH Terms: conditions — Health Education; COVID-19; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental)
  Interventions: Other: health education intervention
- Control (No Intervention)

INTERVENTIONS:
Other: health education intervention — health education intervention
  Arms: Education

SUMMARY:
we aimed to assess the impact of health education on the anxiety level of COVID-19 patients during the isolation period.

DETAILED DESCRIPTION:
This is a randomized controlled trial conducted between February 2021 and June 2021. Patients tested positive for Covid-19 with mild to moderate forms were randomized to Education (n=267) or control (n=269). The education group received a phone health education session on day 1 (D1) following the diagnosis. The three components of the health education intervention were an explanation of the coronavirus disease, what to do in the event of complications, and the recommended preventive measures. The two groups received a telephone evaluation of their Hospital Anxiety and Depression scores on (D1) and day seven D7 following the positive diagnosis. The primary outcome was the rate of anxiety reduction in each group at D7 based on a HAD-A score ≥ 8. Secondary outcomes were the rate of anxiety reduction at D7 based on a HAD-A score ≥ 11, the percentage of people complying with isolation and the scores of adherence to preventive measures during the isolation in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Covid-19 after positive PCR or positive antigen rapid test, over 18 years of age, who did not require hospitalization

Exclusion Criteria:

* Patients not reachable at the first day phone call of the diagnosis and patients unable to answer the telephone questionnaire due to their cognitive state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
The rate of anxiety reduction | One week (7 days) after the COVID 19 diagnosis
  The rate of anxiety reduction in each group at Day 7 based on a HAD-A score ≥ 8

CONTACTS AND LOCATIONS:
Locations (1):
- Fattouma Bourguiba University Hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zemni I, Gara A, Nasraoui H, Kacem M, Maatouk A, Trimeche O, Abroug H, Fredj MB, Bennasrallah C, Dhouib W, Bouanene I, Belguith AS. The effectiveness of a health education intervention to reduce anxiety in quarantined COVID-19 patients: a randomized controlled trial. BMC Public Health. 2023 Jun 20;23(1):1188. doi: 10.1186/s12889-023-16104-w. PMID 37340300